CLINICAL TRIAL: NCT02642237
Title: The Effects of an Endotoxin Challenge on the Immune Response Elicited by a Subsequent Challenge With Fluenz in Healthy Volunteers, an Explorative Study
Brief Title: The Effects of Preceding LPS Administration on the Fluenz-induced Immune Response
Acronym: LPS-Fluenz
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Principal Investigator, Matthijs Kox, Principal investigator, Radboud University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: LPS-Fluenz
Record Dates: First submitted 2015-12-14; First posted 2015-12-30 (Estimated); Results first posted 2019-04-19 (Actual); Last update posted 2019-05-14 (Actual); Status verified 2019-05

CONDITIONS: Innate Immune Response; Immune Tolerance
Keywords: Fluenz; innate immune response; endotoxin tolerance; priming

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LPS-Fluenz (Experimental): Healthy volunteers administered intravenously with endotoxin, followed by an intranasal inoculation with Fluenz, a live-attenuated influenza vaccin
  Interventions: Biological: Fluenz; Other: LPS
- Placebo-Fluenz (Placebo Comparator): Healthy volunteers administered intravenously with placebo, followed by an intranasal inoculation with Fluenz, a live-attenuated influenza vaccin
  Interventions: Biological: Fluenz; Other: placebo

INTERVENTIONS:
Biological: Fluenz — intranasal inoculation with Fluenz
Other: placebo
  Arms: Placebo-Fluenz
Other: LPS
  Arms: LPS-Fluenz

SUMMARY:
To evaluate the bacterial-viral interactions between LPS and Fluenz as a model for sepsis (bacterial) and Influenza (viral) infections which are common and associated with high mortality rates in the ICU. To understand these interactions is important for the development of preventive and therapeutic interventions.

DETAILED DESCRIPTION:
The Influenza virus is known for its severe course of infection and systemic effects, associated with high mortality rates. Recent work has shown that influenza promotes susceptibility for secondary bacterial infections, thereby worsening the prognosis. While it has become clear that bacterial infections induce an immunosuppressed state in which the immune response against viral infections is attenuated1, it is unknown how a bacterial infection, such as in sepsis, influences the susceptibility and immune response to influenza. The sepsis-induced immunosuppressive state, called "immunoparalysis", may be a major contributor to this increased vulnerability. Because of the high mortality rates of both sepsis and influenza, it is of main importance to understand this interaction for the development of putative preventive and therapeutic interventions in ICU patients.

Human endotoxemia represents a model of systemic inflammation, mimicking bacterial sepsis and subsequent development of immunoparalysis. The live, attenuated, quadrivalent influenza vaccine "Fluenz™" is registered in the European Union and can be used as a surrogate for an actual influenza infection. In this study, we want to investigate the effects of an endotoxemia challenge on the Fluenz™-induced inflammatory response to present unique in vivo data on mechanistic interactions of systemic LPS followed by mucosal Fluenz™, thereby providing clues regarding the increased vulnerability towards viral infections in septic patients and open up new avenues to investigate therapeutic measures to prevent this. Furthermore, it provides important implications regarding the safety and efficacy of the vaccine in (post)septic or immunocompromised patients.

Objective: Our primary objective is to investigate the effects of endotoxin-induced systemic inflammation and subsequent development of endotoxin tolerance on the inflammatory response following Fluenz administration in vivo. To evaluate whether these effects involve local and/or systemic inflammation, symptoms, temperature and peak expiratory flow will be measured. Next, local inflammatory parameters are measured in nasal wash and systemic inflammatory parameters are measured in blood. Furthermore, we want to evaluate whether preceding endotoxemia influences the viral shedding of influenza in nasal wash. Also, changes in the mucosal microbiome, transcriptome and metabolome will be assessed. Finally, mitochondrial function and mental strength during human endotoxemia will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy

Exclusion Criteria:

* Pre-existent lung disease, including asthma, severe allergic rhinitis
* Use of any medication
* Current smoker or more than 5 pack-year history
* Use of recreational drugs within 21 days prior to start of the study
* Use of caffeine or alcohol within 1 day prior to start of the study
* Surgery or trauma with significant blood loss or blood donation within 3 months prior to start of the study
* Participation in another clinical trial within 3 months prior to start of the study
* Frequent nosebleeds
* Recent nasal or otologic surgery
* (suspected) influenza infection during the last year
* Clinically significant acute (febrile) illness or a common cold within four weeks prior to start of the study
* History of frequent vaso-vagal collapse or of orthostatic hypotension History, signs or symptoms of cardiovascular disease.
* History of allergic reaction to Fluenz™, eggs / gelatin / gentamicin
* History of Guillain-Barré Syndrome
* Cardiac conduction abnormalities on the ECG consisting of a 2nd degree atrioventricular block or a complex bundle branch block.
* Hypertension (defined as Blood pressure (RR) systolic > 160 or RR diastolic > 90).
* Hypotension (defined as RR systolic < 100 or RR diastolic < 50).
* Renal impairment (defined as plasma creatinin >120 μmol/l).
* Liver function abnormality: alkaline phosphatase>230 U/L and/or Alanine-aminotransferase (ALT)>90 units per Liter (U/L)
* C-reactive protein (CRP) > 20 mg/L, white blood cell count (WBC) > 12x109/L
* Vaccination with influenza this season
* Recent vaccination

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2018-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Pickkers, Prof. Dr., Principal Investigator — Radboud University Medical Center

RESULTS

PARTICIPANT FLOW:
Groups:
- LPS-Fluenz: Healthy volunteers administered intravenously with endotoxin, followed by an intranasal inoculation with Fluenz, a live-attenuated influenza vaccin
  Fluenz: intranasal inoculation with Fluenz
  LPS
- Placebo-Fluenz: Healthy volunteers administered intravenously with placebo, followed by an intranasal inoculation with Fluenz, a live-attenuated influenza vaccin
  Fluenz: intranasal inoculation with Fluenz
  placebo
Period: Overall Study
Arm/Group | LPS-Fluenz | Placebo-Fluenz
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LPS-Fluenz | Placebo-Fluenz | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 15 | 30
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 15 | 15 | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 15 | 15 | 30
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Netherlands | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Peak Levels of Interferon Gamma-induced Protein 10 (IP-10) in Nasal Wash Fluid
Description: Interferon gamma-induced protein 10 is a marker of viral-induced inflammation. Higher levels indicate a more pronounced inflammatory response upon a viral infection.
Time Frame: 35 days after FLuenz inoculation
Measure: Geometric Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | LPS-Fluenz | Placebo-Fluenz
Number analyzed (Participants) | 15 | 15
pg/mL | 2000 [900 to 3000] | 1900 [900 to 2800]

ADVERSE EVENTS:
Arm/Group | LPS-Fluenz | Placebo-Fluenz
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No